CLINICAL TRIAL: NCT06140654
Title: Oral Quality of Life and Food Intake Survey
Brief Title: Oral Health-related Patterns of Food Selectivity in Dental Populations
Status: Completed | Type: Observational
Sponsor: Hôpital Rothschild (Other)
Responsible Party: Principal Investigator, Dr Braud Adeline, Professor in oral rehabilitation, Hôpital Rothschild
Other Study IDs: 17-BRAU-02
Record Dates: First submitted 2023-11-14; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-11

CONDITIONS: Oral Disease; Food Selection
Keywords: eating behavior; food preferences
MeSH Terms: conditions — Mouth Diseases; Food Preferences; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-dental group: 62 non-seeking dental treatment subjects, aged 30-65 years, previously recruited within the general population from december 2017 to january 2018. Declared painful conditions including temporo-mandibular disorder, cephalalgia, oral or dental pain were initially considered as excluding conditions. Exclusion criteria also included diagnosis of acute orofacial disease (i.e. rhinitis) or sensory trouble (i.e. anosmia, dysgeusia) neither at the time of the experiment nor in the recent past, pregnancy, head and neck irradiation, eating disorders, enteral or parenteral feeding, and cognitive impairment or impaired communication.
  They took part in an individual session with a dental practitioner of about 30-min during which food selectivity, medical history, and oral health status were assessed.
  Interventions: Diagnostic Test: Clinical oral examination; Diagnostic Test: Food behavior
- Dental group: 63 patients recruited from September 2019 to December 2020 among patients seeking/pending dental treatment within the university dental clinic of the Rothschild hospital (AP-HP Sorbonne University, Paris, France). Inclusion criteria were: age between 35 and 65 years, literate French speakers, willing and able to complete the survey in a single setting. Patients suffering from cognitive impairment or impaired communication were excluded.
  They took part in an individual session with a dental practitioner of about 30-min during which food selectivity, medical history, and oral health status were assessed.
  Interventions: Diagnostic Test: Clinical oral examination; Diagnostic Test: Food behavior

INTERVENTIONS:
Diagnostic Test: Clinical oral examination — Clinical oral examinations are conducted by a dental practitioner. They point out the number of teeth (ranging from 0 to 32), the number of occlusal functional units (OFU, ranging from 0 to 10, with one unit considered as a pair of antagonist premolars and molars that had at least one contact area during maximum intercuspal relationships, evaluated by asking the participants to clench on a 200 µm thick articulating paper, the presence of dental prostheses (fixed prosthesis and removable denture), the number of denture worn during meals (removable partial or complete denture, either maxillary or mandibular, or both, with number ranging from 0 to 2), the number of decayed, missing, filled teeth (DMFT index, based on 28 teeth), and the Russel's periodontal index which is presently preferred to the Community (namely CPITN) because it takes tooth mobility into account.
Diagnostic Test: Food behavior — Food selective behavior is assessed using a food selectivity questionnaire previously developed for French adults 34. Participants will be interviewed and asked to check each food item they do not eat among a list of 71 familiar products which includes raw foods and dishes from the following categories: starters, meat, fish, egg, garnish, dairy products, desserts, bread, and beverages. A food selectivity score corresponding to the total number of avoided foods will be assessed for each participant. For each avoided food, participants explain why they do not eat it among reasons including "I don't know it", "I dislike it", "I suffer from chewing or swallowing it (oral discomfort)", "I experience difficulties digesting the food", "This food is forbidden for medical reason", and "This food is forbidden for ethical or religious reasons".

SUMMARY:
The present study was undertaken in order to describe the clinical profiles of food selective behavior in 35-65 years dental and non-dental populations.

DETAILED DESCRIPTION:
The study population included 125 participants, recruited within the general population and in a dental clinic: -Non-dental group included 62 non-seeking dental treatment subjects, aged 30-65 years, previously recruited during the OralPom survey. -Dental group included 63 patients recruited from September 2019 to December 2020 among patients seeking/pending dental treatment within the university dental clinic of the Rothschild hospital (AP-HP Sorbonne University, Paris, France).

Both groups took part in an individual session with a dental practitioner during which food selectivity, medical history, and oral health status were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Non-dental group : non-seeking dental treatment subjects, aged 30-65 years.
* Dental group: patients seeking/pending dental treatment within the university dental clinic of the Rothschild hospital (AP-HP Sorbonne University, Paris, France), aged between 35 and 65 years, literate French speakers, willing and able to complete the survey in a single setting.

Exclusion Criteria:

* For non dental group :Declared painful conditions including temporo-mandibular disorder, cephalalgia, oral or dental pain, diagnosis of acute orofacial disease (i.e. rhinitis) or sensory trouble (i.e. anosmia, dysgeusia) neither at the time of the experiment nor in the recent past, pregnancy, head and neck irradiation, eating disorders, enteral or parenteral feeding, and cognitive impairment or impaired communication.
* Patients suffering from cognitive impairment or impaired communication are excluded.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French adults, aged from 30 to 65 years old.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Food selectivity score | During clinical examination session (1 hour) at baseline
  The food selectivity score measures the number of avoided foods. The score ranges from 0 to 71, 0 meaning no food selectivity and 71 meaning high food selectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Braud, PhD, Principal Investigator — Unievrsité Paris Cité
Locations (1):
- Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No